CLINICAL TRIAL: NCT07113925
Title: A Phase I Clinical Trial Evaluating the Safety and Efficacy of TQB2101 in Subjects With Advanced Hematologic Malignancies
Brief Title: A Clinical Trial Evaluating TQB2101 in Subjects With Advanced Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2101-I-02
Record Dates: First submitted 2025-07-31; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-04

CONDITIONS: Advanced Hematologic Malignancies
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2101 for Injection (Experimental): Intravenous injection, administered starting on Day 1 of each cycle, with a treatment cycle every 3 weeks; the dose levels range from 0.4 mg/kg to 1.6 mg/kg.
  Interventions: Drug: TQB2101 for Injection

INTERVENTIONS:
Drug: TQB2101 for Injection — TQB2101 for Injection is an ROR1 ADC, an antibody-drug conjugate. It consists of three main components: a ROR1 monoclonal antibody responsible for selectively recognizing the surface antigen of cancer cells, a small molecule toxin responsible for killing cancer cells, and a linker connecting the antibody and the small molecule toxin. It is intended for clinical use in the treatment of advanced malignant tumors, including advanced malignant hematological tumors.

SUMMARY:
TQB2101 for Injection is an Antibody-Drug Conjugate (ADC) targeting Receptor Tyrosine Kinase Like Orphan Receptor 1 (ROR1).It consists of three main components: a ROR1 monoclonal antibody responsible for selectively recognizing the surface antigen of cancer cells, a small molecule toxin responsible for killing cancer cells, and a linker connecting the antibody and the small molecule toxin. It is intended for clinical use in the treatment of advanced malignant tumors, including advanced malignant hematological tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in this study, sign the informed consent form, and demonstrate good compliance.
* Age between 18 and 75 years (calculated based on the date of signing the informed consent form).
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
* Expected survival >12 weeks.
* Subjects with advanced hematologic malignancies confirmed by cytology/histopathology, who have failed standard treatment or lack effective treatment options.
* At least one measurable lesion according to the 2014 Lugano criteria: lymph node lesions with long axis >15mm or extranodal lesions with long axis >10mm on CT cross-sectional imaging.
* Adequate organ function meeting the following criteria:

  1. Hemoglobin (HGB) ≥80g/L
  2. Absolute neutrophil count (ANC) ≥1.0×10⁹/L
  3. Platelet count (PLT) ≥75×10⁹/L (≥50×10⁹/L if with bone marrow involvement)
  4. Total bilirubin (TBIL) ≤1.5×ULN
  5. Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤2.5×ULN (≤5×ULN if with liver metastases)
  6. Serum creatinine (CR) ≤1.5×ULN OR creatinine clearance rate (CCR) ≥60ml/min (calculated using standard Cockcroft-Gault formula)
  7. Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT), and International Normalized Ratio (INR) ≤1.5×ULN (without anticoagulation therapy)
* Women of childbearing potential must agree to use effective contraception during the study and for 6 months after study completion, with negative blood pregnancy test within 7 days prior to enrollment; male subjects must agree to use effective contraception during the study and for 6 months after study completion.

Exclusion Criteria:

* Patients with other malignant tumors that occurred within 3 years before the first administration or currently coexisting with other malignant tumors are excluded, except for those who have undergone a single surgical treatment for other malignant tumors and have achieved a disease-free survival (DFS) of 5 consecutive years; patients with cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor invading the basement membrane)] are eligible for inclusion.
* Tumor-related symptoms and treatments:

  1. Lymphoma involving or suspected to involve the central nervous system, or primary central nervous system lymphoma;
  2. Patients who have received chemotherapy, immunotherapy within 4 weeks before the first administration, radiotherapy or small molecule targeted drugs within 2 weeks, or are still within 5 half-lives of the drug (whichever occurs earlier), with a washout period calculated from the end of the last treatment;
  3. Patients who have received treatment with traditional Chinese medicine with clear anti-tumor indications in the National Medical Products Administration (NMPA) approved drug instructions (including Compound Cantharidin Capsules, Kang'ai Injection, Kanglaite Capsules/Injection, Aidi Injection, Brucea javanica Oil Injection/Capsules, Xiaoaiping Tablets/Injection, Huachansu Capsules, etc.) within 2 weeks before the first administration;
  4. Patients who have previously received treatment with ROR1 inhibitor drugs;
  5. Patients who have participated in other anti-tumor drug clinical trials within 4 weeks before the first administration (calculated from the last use of the trial drug) and have used the trial drug, or are still within 5 half-lives of the study drug (whichever is shorter).
* Patients with adverse reactions from previous treatments that have not recovered to a Common Terminology Criteria for Adverse Events Version 5.0 (CTC AE v5.0) grade score of ≤1, except for alopecia, non-clinically significant and asymptomatic laboratory abnormalities, and stable hypothyroidism treated with hormone replacement therapy, which are judged by the investigator to have no safety risks.
* Patients who have undergone major surgical treatment, significant traumatic injury, or are expected to undergo major surgery during the study treatment period (except for surgeries specified in the protocol) within 4 weeks before the first administration, or have long-term unhealed wounds or fractures.
* Patients who have experienced any bleeding event ≥ CTC AE v5.0 grade 3 within 4 weeks before the first administration, or have bleeding or coagulation disorders and are using warfarin, aspirin, or other antiplatelet aggregation drugs (except for maintenance doses: aspirin ≤ 100mg/d, clopidogrel ≤ 75mg/d), or have any bleeding signs or history judged by the investigator to be unsuitable for inclusion.
* Patients who have experienced arterial or venous thrombotic events within 6 months before the first administration, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, and pulmonary embolism.
* Patients with decompensated liver cirrhosis (Child-Pugh liver function rating of B or C), active chronic hepatitis B, or active hepatitis C: HbsAg positive and hepatitis B virus (HBV) DNA positive or with a detection value exceeding the lower limit of detection; HCV antibody positive and HCV RNA positive or with a detection value exceeding the lower limit of detection.

Note: For eligible HbsAg positive patients with hepatitis B, regardless of whether HBV DNA is detectable, continuous antiviral treatment (recommended nucleotide analogues) and regular monitoring of HBV DNA are required; for patients with positive HBcAb but negative HbsAg, regular monitoring of HBV DNA is required, and preventive antiviral treatment is recommended; for patients with hepatitis C, regular monitoring of hepatitis C virus (HCV) RNA is required.

* Patients with active syphilis requiring treatment.
* Patients with active pulmonary tuberculosis, a history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonia, radiation pneumonitis requiring treatment, or active pneumonia with clinical symptoms. (10) Subjects with a history of substance abuse of psychotropic drugs and unable to quit or with mental disorders.
* Subjects with a history of decompensated liver cirrhosis and hepatic encephalopathy.
* Subjects with clinically significant cardiovascular diseases, including any of the following conditions:

  1. Subjects who have experienced acute myocardial infarction or severe/unstable angina within 6 months before the start of study treatment; or subjects with New York Heart Association (NYHA) functional classification of grade 2 or higher heart failure;
  2. Subjects with prolonged QT interval corrected by the Fridericia formula (QTcF) at rest, with QTc ≥ 450 ms (male) or QTc ≥ 470 ms (female);
  3. Subjects with a history of or ongoing severe uncontrolled ventricular arrhythmias requiring drug treatment;
  4. Left ventricular ejection fraction (LVEF) < 50%;
  5. Congenital long QT syndrome or any known history of torsades de pointes (TdP);
  6. Uncontrolled hypertension (after standard antihypertensive treatment, systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 90 mmHg), or a history of hypertensive encephalopathy/hypertensive crisis.
* Subjects with active or uncontrolled severe infections (≥ CTC AE v5.0 grade 2 infection).
* Subjects with renal failure requiring hemodialysis or peritoneal dialysis.
* Subjects with a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases.
* Subjects with (non-infectious) pneumonia/interstitial lung disease requiring steroid treatment or currently having non-infectious pneumonia/interstitial lung disease or having been hospitalized or treated with therapeutic antibiotics for any active infection within 4 weeks before the start of study treatment, including but not limited to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection.
* Subjects with a history of or current central nervous system diseases, including but not limited to epilepsy, hemorrhagic/ischemic stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, paralysis, aphasia, mental disorders, consciousness disorders, unexplained coma, neuropathy, organic brain syndrome, etc.; and subjects who have experienced cerebrovascular accidents, cerebral infarction, etc. within 6 months before the first dose.
* Subjects with urine protein ≥ ++ in routine urine test and confirmed 24-hour urine protein quantification > 1.0 g.
* Poorly controlled diabetes (fasting blood glucose (FBG) > 10 mmol/L).
* Uncontrolled pleural, peritoneal or pericardial effusion requiring repeated drainage or with obvious symptoms. Subjects with only a small amount of pleural effusion, ascites or pericardial effusion shown on imaging, without symptoms and without drainage or other treatment within 2 weeks before enrollment, can be enrolled.
* Subjects known to be allergic to the excipients of the study drug.
* Subjects, as judged by the investigator, with conditions that seriously endanger the safety of the subject or affect the subject's ability to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Up to 24 months
  Dose-limiting toxicity (DLT) refers to any Grade 3-5 adverse event (as per National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0) considered related to the investigational drug and occurring from the first dose administration through the end of the first treatment cycle.
Maximum Tolerated Dose | Up to 24 months
  Defined as the highest dose in less than 33% of subjects with dose-limiting toxicity (DLT).
Phase II recommended dose | Up to 24 months
  The recommended dose for subsequent phase II studies will be determined based on Maximum Tolerated Dose, Pharmacokinetics, preliminary efficacy and safety.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 24 months
  Proportion of subjects achieving best overall response of PR or CR.
Disease Control Rate (DCR) | Up to 24 months
  Proportion of subjects achieving best overall response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD).
Progression-Free Survival (PFS) | Up to 24 months
  The time from the first dose of the investigational drug to the first documented disease progression or death (from any cause), whichever occurs earlier.
Overall Survival (OS) | Up to 24 months
  The time from the first dose of the investigational drug to the date of death due to any cause.
Incidence and severity of adverse events (AEs) | Up to 24 months
  Incidence and severity of adverse events (AEs)
Incidence and severity of laboratory abnormalities | Up to 24 months
  Incidence and severity of laboratory abnormalities
Incidence and severity of serious adverse events (SAEs) | Up to 24 months
  Incidence and severity of serious adverse events (SAEs)
Incidence of anti-drug antibodies (ADA) | Up to 24 months
  Incidence of anti-drug antibodies (ADA)
Total antibody (TA) | Up to 6 cycles, ecah cycle is 21 days
  Total antibody (TA)
Total antibody-drug conjugate (ADC) | Up to 6 cycles, ecah cycle is 21 days
  Total antibody-drug conjugate (ADC)
Total small-molecule toxin (SMT) | Up to 6 cycles, ecah cycle is 21 days
  Total small-molecule toxin (SMT)

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality